CLINICAL TRIAL: NCT00053742
Title: A Phase I/II Clinical Trial of Modified Vaccinia Virus Ankara (MVA) to Evaluate Its Safety, Immunogenicity and Protective Efficacy Against Dryvax® (Registered Trademark) Challenge in Vaccinia-Immune Individuals
Brief Title: Phase I/II Trial of Modified Vaccinia Virus Ankara (MVA) Vaccine Against Smallpox
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 030087; 03-I-0087
Record Dates: First submitted 2003-02-04; First posted 2003-02-05 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2006-03

CONDITIONS: Healthy
Keywords: Smallpox; Vaccine; Vaccination; Variola; Adults; Healthy Volunteer; HV; Smallpox Vaccine
MeSH Terms: conditions — Smallpox

INTERVENTIONS:
Drug: Modified Vaccinia Virus Ankara TBC-MVA

SUMMARY:
This study will test the safety of an experimental vaccine called modified vaccinia virus ankara (MVA) and determine if it confers protection against the smallpox virus (variola). There is an existing vaccine, called Dryvax® (Registered Trademark), which is effective against smallpox; however, this vaccine can cause various side effects, including some that, on rare occasions, can be life-threatening. Dryvax® (Registered Trademark) has not been used in the United States since childhood vaccination was stopped in 1971, and though it is given to certain healthcare and laboratory workers, and some people in the armed forces, it is not recommended for the general population. Both the MVA and Dryvax® (Registered Trademark) vaccines are made using the vaccinia virus, which is closely related to variola.

Healthy normal volunteers between 31 and 60 years of age who have been vaccinated with a smallpox vaccine more than 10 years before entering the study may be eligible for this protocol. Candidates will be screened with a medical history, physical examination, and blood and urine tests, including an HIV test and a pregnancy test for women of childbearing potential.

Participants will receive MVA vaccine or placebo, followed by a dose of Dryvax® (Registered Trademark). The MVA vaccine and placebo are injected into an arm muscle with a needle and syringe. The Dryvax® (Registered Trademark) vaccine is administered with a special forked needle that is poked lightly into the skin of the upper arm, usually 15 times, in a process called scarification. When the vaccine works, a small pus-filled blister forms, followed by a scab and then scarring at the site of the vaccination. The formation of the blister and scab is called a take, indicating that the vaccine is effective and will protect against smallpox for at least a few years. If scarification does not take, it can either mean that the person already has immunity or that the vaccine did not work.

Study participants will be randomly assigned to one of the following dosing groups: 1) one injection of MVA; 2) one injection of placebo; 3) two injections of MVA 4 weeks apart; or 4) two injections of placebo 4 weeks apart. All participants will receive a challenge dose of Dryvax® (Registered Trademark) 12 weeks after their last injection of MVA or placebo to determine if the MVA vaccine has conferred immunity. A take, that occurs in response to the Dryvax® (Registered Trademark) dose indicates lack of prior immunity, and thus tells whether one or two doses of MVA is needed to produce an immune response.

Participants will be observed for at least 1 hour after each injection. They will come to the clinic at least once a week after MVA or placebo injections and at least twice a week after Dryvax® (Registered Trademark) to have the injection site evaluated and photographed. At each visit, participants will be asked how they are feeling and what medications, if any, they are taking. Blood and urine tests will be done according to the following schedule:

* Before each injection;
* 1 week after each injection;
* 4 weeks after the MVA or placebo injections are finished;
* At the time of the Dryvax® (Registered Trademark) dose;
* 4 weeks after the Dryvax® (Registered Trademark) dose;
* 12 weeks after the Dryvax® (Registered Trademark) dose.

Additional laboratory tests may be done between visits if medically necessary.

DETAILED DESCRIPTION:
This is a phase I/II, randomized, placebo-controlled, double-blinded, study of MVA vaccine. The hypothesis is that MVA will be safe in vaccinia-immune adults when administered by intramuscular injection, and that this vaccine will result in an immunologic response comparable to that observed after Dryvax® (Registered Trademark) vaccination in previously vaccinia-immunized persons. The primary objectives include: evaluating the safety of MVA administered by intramuscular (IM) injection at 10(8) PFU, and determining whether MVA provides clinical evidence of protection against a 12-week Dryvax challenge when compared to placebo groups. The secondary objectives are to identify the schedules of MVA administration that provide clinical evidence of protection against Dryvax® (Registered Trademark) challenge and compare the Immunogenicity of Dryvax® (Registered Trademark) and MVA as measured by vaccinia-specific neutralizing antibody, ELISA and intracellular cytokine assays, as well as variola-specific neutralizing antibody assays that will be conducted at the CDC on a subset of samples.

ELIGIBILITY:
INCLUSION CRITERIA:

A participant must meet all of the inclusion criteria, as follows:

1. Age born no later than 1979 - age 60 years old
2. Prior vaccination more than 10 years ago with any vaccinia product and evidence of a scar typical of prior vaccination leading to a primary take.
3. Available for follow-up for the duration of the study (at least 28 weeks).
4. Able and willing to sign the informed consent form
5. Willing to allow blood samples to be stored for future research
6. In good general health, without clinically significant medical history, physical examination findings or laboratory results.
7. Hematocrit greater than or equal to 34% for women; greater than or equal to 38% for men
8. White blood cell count within institutional normal limits
9. Differential either within institutional normal range or accompanied by site physician approval
10. Total lymphocyte count greater than or equal to 1000 cells/mm(3)
11. Absolute CD4 count greater than or equal to 400 cells/mm(3)
12. Platelets within institutional normal limits
13. ALT (SGPT) less than or equal to institutional upper normal limit
14. Serum creatinine less than or equal to 1.3 mg/dL and calculated creatinine clearance (CrCl) greater than or equal 55 mL/min using the formula below:

    Male CrCl (mL/min) = [140 - age (yrs)] x [body wt (kg)] / 72 x [serum Cr (mg/dL)]

    Female CrCl (mL/min) = [140 - age (yrs)] x [body wt (kg) x .85] / 72 x [serum Cr (mg/dL)]
15. Normal urinalysis defined as: negative glucose, negative or trace protein, and negative or trace hemoglobin
16. Negative hepatitis B surface antigen (HBsAg)
17. Negative anti-HCV or negative HCV PCR if the anti-HCV is positive
18. Negative HIV ELISA and HIV PCR (volunteers who have previously participated in an HIV vaccine study are eligible with positive ELISA if Western blot is indeterminate or negative and HIV PCR is negative.)
19. Negative serum beta-HCG test for women presumed to be of reproductive potential.
20. A female participant must meet one of the following criteria: a) no reproductive potential due to menopause (one year without menses), hysterectomy, bilateral oophorectomy, or tubal ligation; b) agrees to consistently practice contraception at least 30 days prior to enrollment and throughout the duration of the study by means of IUD, hormone-based therapy (e.g., contraceptive pills, Norplant (Registered Trademark), or Depo-Provera (Registered Trademark)) or other FDA-licensed methods).
21. Able to provide proof of identity to the acceptance of the study clinician completing the enrollment process.

EXCLUSION CRITERIA:

Volunteers are excluded from study participation if one or more of the following is true:

1. Vaccination with any vaccinia product within the last 10 years including vaccination with any vaccinia recombinant product.
2. Diseases or conditions that cause immunodeficiency (examples are HIV AIDS, leukemia, lymphoma, generalized malignancy, agammaglobulinemia, history of transplantation, or therapy with alkylating agents, antimetabolites, radiation, or oral or parental corticosteroids).
3. In close physical contact (household or at work) with an individual who has the diseases or conditions that cause immunodeficiency.
4. History of eczema, even if the condition is mild or not presently active.
5. In close physical contact (household or at work) with an individual who has eczema, even if mild or not presently active.
6. Acute or chronic skin conditions such as atopic dermatitis, burns, impetigo, or varicella zoster (shingles).
7. Household member who is pregnant.
8. Women who are breast-feeding.
9. Household member less than 1 year old or work with children less than 1 year old.
10. Serious, life-threatening allergies to antibiotics polymixin B, streptomycin, tetracycline, neomycin or cidofovir.
11. Allergy to eggs or blood products (including Immunoglobulin products) or hypersensitivity to probenicid or sulfa-containing medications.
12. Receipt of live attenuated viruses within 30 days prior to enrollment.
13. Receipt of subunit or killed vaccines within 14 days prior to enrollment.
14. Use of investigational research agents within 30 days prior to enrollment.
15. Receipt of blood products within 120 days prior to HIV screening.
16. Receipt of immunoglobulin within 60 days prior to HIV screening.
17. History of serious adverse reactions to vaccines, such as anaphylaxis and related symptoms such as hives, respiratory difficulty, angioedema and abdominal pain.
18. History of type I or type II diabetes mellitus, except gestational diabetes or diabetes controlled with diet alone.
19. Currently taking anti-TB prophylaxis or therapy.
20. History of seizure disorder other than: a) febrile seizures under the age of two, or b) seizures secondary to alcohol withdrawal more than 3 years ago, or c) a singular seizure more than 3 years ago.
21. Bleeding disorder that was diagnosed by a physician, (e.g., factor deficiency, coagulopathy, or platelet disorder that requires special precautions).
22. Splenectomy.
23. Hypertension that is not well controlled by medication or is more than 150/100 at enrollment.
24. Psychiatric condition that precludes compliance with the protocol; past or present psychoses; past or present bipolar disorder requiring therapy that has not been well-controlled on medication within the past two years; disorder requiring lithium; suicidal ideation occurring within five years prior to enrollment.
25. Any medical, psychiatric, social condition, or occupational or other responsibility that, in the judgement of the investigator, would interfere with or serve as a contraindication to adherence to the study protocol or ability to give informed consent.
26. History of cardiomyopathy, myocardial infarction, angina, congestive heart failure, coronary artery disease, stroke, transient ischemic attack, or history of 3 or more risk factors for coronary heart disease from the following list:

current cigarette smoking;

high blood pressure diagnosed by a doctor;

high blood cholesterol diagnosed by a dicotr or a fasting LDL greater than 160 mg/dL at screening;

diabetes diagnosed by a doctor;

a first-degree relative (father, mother, brother, sister) who had coronary artery disease before the age of 50.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 80
Dates: Start 2003-02; Study Completion 2006-03

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Allergy and Infectious Diseases (NIAID), Bethesda, Maryland, United States

REFERENCES:
- [Background] Stittelaar KJ, Osterhaus AD. MVA: a cuckoo in the vaccine nest? Vaccine. 2001 Jun 14;19(27):V-VI. doi: 10.1016/s0264-410x(01)00171-2. No abstract available. PMID 11395217
- [Background] Henderson DA, Inglesby TV, Bartlett JG, Ascher MS, Eitzen E, Jahrling PB, Hauer J, Layton M, McDade J, Osterholm MT, O'Toole T, Parker G, Perl T, Russell PK, Tonat K. Smallpox as a biological weapon: medical and public health management. Working Group on Civilian Biodefense. JAMA. 1999 Jun 9;281(22):2127-37. doi: 10.1001/jama.281.22.2127. PMID 10367824
- [Background] Henderson DA. The looming threat of bioterrorism. Science. 1999 Feb 26;283(5406):1279-82. doi: 10.1126/science.283.5406.1279. PMID 10037590